CLINICAL TRIAL: NCT02191150
Title: Retrospective Study of Stable Haemodialysis Patients Switched From Darbepoetin Alfa to Epoetin Alfa Biosimilar
Brief Title: Study of Haemodialysis Patients Switching From Aranesp to Biosimilar
Acronym: SHADE
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20130300
Record Dates: First submitted 2014-07-07; First posted 2014-07-16 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Anaemia
Keywords: Anaemia, Chronic Kidney Disease, Switching, Aranesp, Darbepoetin Alfa, Epoetin Alfa Biosimilars, Haemodialysis.
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with CKD

SUMMARY:
The study will obtain data to show insight into clinical outcomes of patients switching from Darbepoetin Alfa to a epoetin alfa biosimilar.

DETAILED DESCRIPTION:
Biosimilars were approved in 2007 by the EMA in EU and in 2010 by the TGA in Australia. This study will look at the retrospective data of patients that have switched from Darbepoetin Alfa to an approved epoetin alfa biosimilar. Data will be collected for the 26 week period prior to switch and a 26 week period post switch to a biosimilar. Data to be collected includes haemoglobin measurements, dose requirements, iron use, any transfusions, hospitalisations and other lab values including TSAT, Ferritin and albumin. Data from the study will be published.

ELIGIBILITY:
Inclusion Criteria

* Patients ≥18 years of age
* Patients with CKD on haemodialysis and fulfilling the following:

  * Received HD for at least 26 weeks prior to switching from treatment with darbepoetin alfa to treatment with an EMA/TGA-approved epoetin alfa biosimilar
  * Received darbepoetin alfa treatment i.v. for at least 26 weeks immediately prior to switching to an EMA/TGA-approved epoetin alfa biosimilar (breaks due to treatment being intentionally withheld are permitted)
  * Switched from darbepoetin alfa treatment to an EMA/TGA-approved epoetin alfa biosimilar at least 26 weeks prior to enrolment
  * Received at least one dose of an EMA/TGA-approved epoetin alfa biosimilar after switching from darbepoetin alfa treatment
* Mean monthly Hb 10-12g/dL in the 12 weeks prior to switch
* Stable darbepoetin alfa dose (i.e. no more than one increment or decrement of PFS) in the 12 weeks prior to switch
* Patient or patient's legally acceptable representative has provided informed consent, if applicable according to local requirements

Exclusion Criteria:

* Treatment with an ESA other than darbepoetin alfa during the 12 weeks prior to switch to biosimilar
* More than 14 days' cumulative treatment with short-acting ESA during weeks 26-13 prior to switch to biosimilar
* Subject received chemotherapy or major surgery during the 26 weeks prior to switch to biosimilar
* Subject was enrolled in an interventional device or drug study at any time during the 52-week data observation period or within 30 days prior to commencement of the data observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises prevalent haemodialysis (HD) patients treated at EU and Australian dialysis clinics after September 2008. Eligible patients will have received treatment with darbepoetin alfa for at least 26 weeks prior to being converted to an EMA/TGA-approved epoetin alfa biosimilar. At each participating study site, all potentially eligible patients are to be considered for enrolment.
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Haemoglobin Concentration | Duration of observation period -52 weeks
  Mean haemoglobin concentration over time

SECONDARY OUTCOMES:
ESA Doses | Duration of observation period -52 weeks
  Doses of ESA over time.
Dose ratio | Start post-switch (weeks 1-4) and pre-switch (weeks -4--1)
  Dose ratio between the start of the post-switch observation period and pre-switch
Dose ratio | Between end of post-switch (weeks 23-26) and pre-switch (weeks -4--1)
  Dose ratio between the end of the post-switch observation period and pre-switch
Haemoglobin excursions | Duration of observation period -52 weeks
  Haemoglobin excursions (<10/dL and >12g/dL)
Haemglobin within range | Duration of observation period -52 weeks
  Haemoglobin in the range 10-12g/dL over time
TSAT, ferritin and albumin values | Duration of observation period -52 weeks
  TSAT, ferritin and albumin over time
Iron Use | Duration of observation period -52 weeks
  Iron use (dose/route) over time
Red cell transfusions (including number of units transfused) | Duration of observation period -52 weeks
  Red cell transfusions (including number of units transfused)
Hospitalisations (including primary cause) | Duration of observation period -52 weeks
  Hospitalisations (including primary cause)

OTHER OUTCOMES:
Number of Subjects with PRCA testing and incidence of neutralizing anti-erythropoietin antibodies | Duration of 52-week observation period
  Pure Red Cell Aplasia (PRCA) test and results

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- Australia (3):
  - Research Site, Herston, Queensland
  - Research Site, Nambour, Queensland
  - Research Site, Woolloongabba, Queensland
- Research Site, Burgas, Bulgaria
- Germany (3):
  - Research Site, Lemgo
  - Research Site, Lich
  - Research Site, Minden
- Greece (5):
  - Research Site, Aigáleo
  - Research Site, Egaleo, Athens
  - Research Site, Kallithea, Athens
  - Research Site, Larissa
  - Research Site, Pátrai
- Italy (2):
  - Research Site, Milazzo ME
  - Research Site, Pisa
- Poland (6):
  - Research Site, Chojnice
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Rybnik
- Spain (2):
  - Research Site, Jaén, Andalusia
  - Research Site, Zamora, Castille and León

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com